CLINICAL TRIAL: NCT05619770
Title: A Single Arm, Open Label, Single Dose and Multiple Dose Study to Evaluate Pharmacokinetics, Safety & Tolerability of 101-PGC-005 in Healthy, Adult, Human Subjects
Brief Title: Study to Evaluate Pharmacokinetics, Safety & Tolerability of 101-PGC-005 in Healthy, Adult, Human Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: 101 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC-005-IN-101
Record Dates: First submitted 2022-11-03; First posted 2022-11-17 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Glucocorticoids Toxicity; COVID-19; Infectious Disease; Virus Diseases
MeSH Terms: conditions — COVID-19; Communicable Diseases; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 101-PGC-005 (Intervention arm) (Experimental): Bolus Injection containing 30mg of 101-PGC-005 will administered intravenously once daily for 3 consecutive days
  Interventions: Drug: 101-PGC-005

INTERVENTIONS:
Drug: 101-PGC-005 — Bolus Injection containing 30mg of 101-PGC-005 will administered intravenously once daily for 3 consecutive days

SUMMARY:
The goal of this interventional study is to evaluate the pharmacokinetics, safety, and tolerability of 101-PGC-005 in healthy, adult, human subjects. The main question it aims to answer is what are the single and multi-dose PK properties of 101-PGC-005 in the systemic circulation

Participants will receive a bolus injection of 101-PGC-005 administered intravenously once daily for 3 consecutive days. Blood and urine samples will be collected at predetermined timepoints for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide audio-visual & written informed consent for participation in the study, and an ability to comprehend the nature and purpose of the study.
* Willing to be available for the entire study period and to comply with protocol requirements. Should have reliable access to the clinical trial center and be available in the area for at least one month.
* Normal, healthy, adult, human subject of 18-45 years (both inclusive) of age.
* Body mass index in the range of 18 -30 kg/m2 (both inclusive).
* Healthy volunteers who are clinically non-anemic will be included as per the discretion of PI/CI/Physician.
* Non-diabetic healthy adult with HbA1c < 5.5 at the time of study entry
* Normal health status as determined by baseline medical and medication history, at the time of screening and vital signs (blood pressure, pulse rate, respiratory rate, and axillary temperature) measurements and physical examination at the time screening as well as check-in during each study period.
* With normal or clinically non-significant laboratory values as determined by hematological, biochemistry tests and urine analysis (included in section no. 9.1).
* With a normal or clinically non-significant 12-lead ECG.
* With a negative test for Human Immunodeficiency Virus (HIV) type I/II antibodies or Hepatitis B surface antigen (HBsAg) or Hepatitis C virus antibodies.
* Non-smokers and should not have been consuming any kind of tobacco products including chewing or inhaling tobacco in the form of jarda, pan, gutkha etc, Or, In case of smokers, they should be willing to abstain from smoking or chewing any tobacco containing product for at least 72.00 hours prior to check-in and throughout the duration of the study till safety samples are collected at the end of the study.
* In case of female subjects:

  * Negative urine pregnancy test during screening and negative serum β- hCG test at check-in.
  * Female subjects with childbearing potential must either abstain from sexual intercourse or use acceptable methods of birth control for at least 15 days before 1st dose till 15 days post last-dose/ entire study period [Acceptable birth control methods include barrier methods such as diaphragm/condom with or without spermicide or who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy has been performed)].
  * They should not be menstruating on the day of the withdrawal of blood, when blood is collected for the purpose of study. Ability to communicate effectively.

Exclusion Criteria:

* History of allergy or hypersensitivity intolerance to Dexamethasone or its formulation excipients which, in the opinion of the clinical investigator, would compromise the safety of the subject or the study.
* Has consumed dexamethasone or any other corticosteroid oral or intravenous for any reasons in past 4 weeks before study entry.
* Hemoglobin level less than 12.5 grams per deciliter for men and 12 grams per deciliter for women.
* Any medical or surgical conditions, which might significantly interfere with the normal functioning of the body or blood forming organs.
* History of severe infection or major surgery in the past 6 months.
* History of Minor surgery or fracture within the past 3 months.
* Significant history or current evidence of malignancy or chronic - infectious, cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic (endocrine), hematological, gastrointestinal, immunological or psychiatric diseases, or organ dysfunction.
* Any major illness or hospitalized within 90 days prior to check-in.
* Any other clinical condition like diarrhea or vomiting within three days prior to dosing.
* Subjects who have been on an unusual or abnormal diet, for whatever reason e.g. because of fasting due to religious reasons during the four weeks before screening.
* Use of any depot injection or an implant of any drug within three months prior to dosing and throughout the study periods.
* Use of any prescribed medication (including herbal medicines and vitamin supplements) within 14 days or within five half-lives of the drug, whichever is longer prior to dosing and throughout the duration of the study until the post study safety sample is collected.
* Use of any OTC products within 7 days or within five half-lives of the drug, whichever is longer prior to first check-in and throughout the duration of the study until the post study safety sample is collected.
* History or presence of gastric or duodenal ulcer or GI bleeding or blood in stools anytime in the past.
* Use of any recreational drug or history of drug addiction.
* Participated in any clinical investigation requiring repeated blood sampling, blood donation, or have blood loss of >300 mL in past 90 days prior to dosing.
* Participated in any clinical study within the past 90 days prior to check-in.
* Use of any Investigational vaccine within the last three years except for Covid-19 vaccines.
* History of Chronic systemic immunosuppressive medications usage for any reasons.
* Consumption of alcohol or alcoholic products within 72.00 hrs prior to dosing in each study period and throughout sampling time points.
* Positive alcohol breath or urine screen for drug of abuse tests during check-in study period.

  > Positive test for alcohol in breath, or drugs of abuse (including benzodiazepines, amphetamines, barbiturates, cocaine, methadone, phencyclidine, 3,4-methylenedioxymethamphetamine [MDMA/ecstasy], tetrahydrocannabinol, and opiates) in urine.
* Consumption of xanthine or its derivative containing food or beverages (e.g. chocolates, tea, coffee or cola drinks) within 48.00 hours prior to dosing in each study period and throughout sampling time points.
* Lactating or nursing female subjects.
* Female subjects using hormonal contraceptive (either oral/implants).
* Any history of difficulty in blood sampling or any vasovagal attack during blood sampling which in the opinion of the Investigator may relevantly interfere with the study sampling.
* Evidence of an uncooperative attitude.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-29 (Actual); Primary Completion 2022-11-03 (Actual); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Single dose PK | -0.5, 0.5, 0.75, 1, 1.5, 2, 3, 6, 9, 12, 24 hours post-dose
  Quantification of 101-PGC-005 concentration available in
  systemic circulation (blood/plasma) in all recruited subjects; pre- and post- dosing with 101-PGC-005 injection on Day 1.
Multiple dose PK | -0.5, 0.5, 0.75, 1, 1.5, 2, 3, 6, 9, 12, 24 hours post-dose
  Quantification of 101-PGC-005 concentration available in systemic circulation (blood/plasma) in all recruited subjects; pre- and post- dosing with 101-PGC-005 injection on Day 3.

SECONDARY OUTCOMES:
Evaluate free dexamethasone levels | -0.5, 0.5, 0.75, 1, 1.5, 2, 3, 6, 9, 12, 24 hours post-dose
  To evaluate free dexamethasone levels available in systemic circulation (blood/plasma) in all recruited subjects; pre- and post- dosing with 101- PGC-005 injection on Day 1 & Day 3.
Evaluate steroid induced hyperglycemia | 5 days
  To evaluate the incidence of steroid-induced hyperglycemia events after 101-PGC-005 administration

OTHER OUTCOMES:
Concentration of 101-PGC-005 in Urine | 0-4, 4-8, 8-12, 12-18, 18-24 hours post-dose
  To evaluate the concentration of unchanged 101-PGC-005 excreted in urine samples of healthy adult subjects after dosing on Day 1.

CONTACTS AND LOCATIONS:
Locations (1):
- ICBio Clinical Research Pvt. Ltd., Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No